CLINICAL TRIAL: NCT01187979
Title: A Proof of Concept Cluster Randomised Controlled Trial to Evaluate the Impact of a Cash Incentivised Prevention Intervention to Reduce HIV Infection in High School Learners in Rural KwaZulu-Natal, South Africa
Brief Title: Reducing HIV in Adolescents
Acronym: RHIVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: MIET Africa (Unknown); KwaZulu-Natal Department of Education (Unknown); Embassy of the Kingdom of the Netherlands (EKN) (Unknown)
Responsible Party: Principal Investigator, Dr Quarraisha Abdool Karim, Principal Investigator and Protocol Chair, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CAPRISA 007
Record Dates: First submitted 2010-08-12; First posted 2010-08-25 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: HIV Infections
Keywords: Cash incentive; HIV prevention; Adolescents; South Africa; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): All eligibly enrolled learners in the intervention schools will receive a prevention program delivered by MIET Africa and the KwaZulu-Natal Department of Education. No cash incentives will be paid for meeting milestones
  Interventions: Behavioral: Life skills curriculum
- Cash incentive (Experimental): All eligibly enrolled learners in the intervention schools will receive a cash incentivised prevention program delivered by MIET Africa and the KwaZulu-Natal Department of Education
  Interventions: Behavioral: Cash incentives; Behavioral: Life skills curriculum

INTERVENTIONS:
Behavioral: Cash incentives — Cash incentives paid to learners for reaching pre-determined milestones
  Arms: Cash incentive
Behavioral: Life skills curriculum — Standard department of education lifeskills curriculum

SUMMARY:
The purpose of this study is to assess the impact of a cash-incentivised prevention intervention on reducing HIV incidence rates in high-school learners in rural KwaZulu-Natal.

DETAILED DESCRIPTION:
The impact of the cash incentivised intervention will be assessed using a matched pair, cluster randomised controlled trial design. The 14 selected high schools in the Vulindlela School Circuit will be matched in pairs. The matched pairs of schools will be the unit of randomisation. Baseline measurements, using a standardised tool (structured questionnaire and biological specimens) will be undertaken simultaneously in each matched pair and will include all eligibly enrolled and consenting learners in the respective schools. On completion of baseline measurements in each matched pair of schools, the randomisation code for the pair will be revealed and the intervention will be implemented in the intervention school. All schools will receive the same prevention intervention but only the intervention school will receive the cash incentives. Follow-up measurements will be undertaken approximately 12 and 24 months after implementation of the intervention using a similar standardised assessment tool to that used at baseline. At baseline and during follow-up assessments in intervention and control schools, linked HIV and substance use testing will be undertaken in all learners and pregnancy testing in female learners. Other secondary endpoints will be assessed using a structured questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Learners must meet all of the following criteria at enrolment in order to be eligible for inclusion in the study:

* Male or female learner in Grade 9 or 10 in one of the 14 selected schools
* Willing and able to provide informed consent and/or assent to participate in the study
* Willing to provide locator data for home visits if necessary
* Not planning to move to another school or relocate in the next 36 months
* Willing to be finger-printed to verify identity for study procedure purposes
* Willing to participate in this study
* Willing to complete all study procedures

Exclusion Criteria:

* Refusal by the learner and/or parent or legal guardian to participate in the study.
* Unable to provide necessary informed consents
* Cognitively challenged learners

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3217 (Actual)
Dates: Start 2010-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
HIV-incidence rates | annually, after every 12 months of follow up
  To evaluate the efficacy of a cash-incentivised prevention intervention in reducing HIV-incidence rates in high-school learners

SECONDARY OUTCOMES:
Academic performance measured as an overall passing grade (50%) | 6 monthly
  To support learners improving academic performance, attend school, complete schooling and improve their self-esteem, learners will be incentivised to pass their June and November examinations, with a minimum of a 50% average. Educators from the selected schools will design, administer and mark the June and November examination papers.
voluntary uptake of HIV testing | annually, after every 12 months of follow up
  Learners must provide the receipt from the clinic that specifies that the learner was tested for HIV.
Substance use patterns | annually, after every 12 months of follow up
  Urine specimens will be utilised for testing for the presence of recreational drugs.
Pregnancy rates in female learners | annually, after every 12 months of follow up
  A dipstick pregnancy test will be performed on the urine sample of all female learners at baseline and at the two annual follow-up visits.
Contraceptive use patterns in female learners | annually, after every 12 months of follow up
  Annual behavioural questionnaires will monitor self-reported contraceptive use.
Participation in extra-curricular activities | annually, after every 12 months of follow up
  Attendance and participation in a life skills/sustainable livelihoods programme will be assessed. Self-reported participation in extra-curricular activities will be assessed in annual behavioural questionnaires.
HIV risk reduction behaviour | Annually, after every 12 months of follow up
  The following will be assessed through a self-reported questionnaire:
  condom use; primary and/or secondary sexual abstinence rates; sexually transmitted disease rates intergenerational sexual coupling (age of sexual partner(s)) age of sexual debut; frequency of HIV testing; number of concurrent sex partners; frequency of partner change; medical male circumcision rates; anal sex rates

CONTACTS AND LOCATIONS:
Overall Officials: Quarraisha Abdool Karim, PhD, Principal Investigator — Associate Scientific Director
Locations (1):
- Vulindlela Clinical Research Site, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pettifor AE, Rees HV, Kleinschmidt I, Steffenson AE, MacPhail C, Hlongwa-Madikizela L, Vermaak K, Padian NS. Young people's sexual health in South Africa: HIV prevalence and sexual behaviors from a nationally representative household survey. AIDS. 2005 Sep 23;19(14):1525-34. doi: 10.1097/01.aids.0000183129.16830.06. PMID 16135907
- [Background] Fernald LC, Hou X, Gertler PJ. Oportunidades program participation and body mass index, blood pressure, and self-reported health in Mexican adults. Prev Chronic Dis. 2008 Jul;5(3):A81. Epub 2008 Jun 15. PMID 18558031
- [Background] Hargreaves JR, Glynn JR. Educational attainment and HIV-1 infection in developing countries: a systematic review. Trop Med Int Health. 2002 Jun;7(6):489-98. doi: 10.1046/j.1365-3156.2002.00889.x. PMID 12031070
- [Derived] Ayton SG, Pavlicova M, Abdool Karim Q. Identification of adolescent girls and young women for targeted HIV prevention: a new risk scoring tool in KwaZulu Natal, South Africa. Sci Rep. 2020 Aug 3;10(1):13017. doi: 10.1038/s41598-020-69842-x. PMID 32747693
- See also: CAPRISA website — http://www.caprisa.org/